CLINICAL TRIAL: NCT01622491
Title: Effectiveness of the GSK Pandemic H1N1 Influenza Vaccines in Preventing Hospitalization for Influenza and Pneumonia in Manitoba, Canada
Brief Title: Effectiveness of H1N1 Influenza Vaccines in Manitoba, Canada
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: International Centre for Infectious Diseases, Canada (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: ICID-2012-H1N1-01
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Influenza; Pneumonia
Keywords: H1N1; pandemic; influenza; pneumonia; vaccine; effectiveness; Manitoba; Canada
MeSH Terms: conditions — Influenza, Human; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Case control: A case-control study with cases (individuals hospitalized with influenza or pneumonia during the second wave of the pandemic) and controls (non-hospitalized individuals) identified using the MH Hospital Separation Abstract Database and the MH Population Registry, respectively. Information on receipt of vaccines will be obtained by record linkage to the MIMS.

SUMMARY:
Excellent immune responses following 1 or 2 doses of the GSK monovalent AS03-adjuvanted pandemic H1N1 (pH1N1) vaccines (e.g., Arepanrix®) have been documented in several trials. Observational studies have found that these vaccines were effective in preventing laboratory confirmed influenza infections. However, it remains unclear whether vaccination during the pandemic was associated with reductions in more clinically meaningful outcomes, such as hospitalizations, severe illness, complications, and death.

The investigators propose to evaluate the effectiveness of the GSK adjuvanted and non-adjuvanted pH1N1 vaccines used in Manitoba in preventing hospitalization and severe illness (defined as illness necessitating admission to intensive care or associated with major complications) due to influenza or pneumonia by means of a case-control study using data from Manitoba Health (MH) administrative databases and the database of the Cadham Provincial Laboratory. The primary outcome will be hospitalization with laboratory-confirmed influenza or pneumonia. A secondary outcome will be hospitalization with influenza or pneumonia. The investigators will also assess the effectiveness of the above vaccines for different age groups and among high-risk populations, e.g., immunocompromised individuals.

DETAILED DESCRIPTION:
Testing for influenza is largely discretionary because most patients presenting with influenza-like illness (ILI) could be effectively and safely managed even when the diagnosis is not confirmed. So, it is unclear whether reduction in the risk of laboratory-confirmed influenza or mild ILI among vaccinated individuals is of much clinical significance. In contrast, hospitalization due to influenza or pneumonia is usually not as discretionary, and from both clinical and public health perspectives avoiding hospitalization is more important and relevant objective for influenza control than the mere reduction of laboratory-confirmed cases.

Thus far there have been few observational studies that examined the effectiveness of the H1N1 vaccine against hospitalization, and most of them had significant limitations including small sample sizes, information limited to certain age groups (e.g., children) and the potential for selection and recall bias. Using data from a Scottish general practice sentinel surveillance network, Simpson et al reported that the adjuvanted GSK vaccine was 95% (76-100%) effective against laboratory-confirmed H1N1 infections, and 100% (∞-100%) effective against hospitalization for influenza and pneumonia. Unexpectedly, the vaccine was equally effective among 'high-risk' groups. Small number of cases limited the precision of these estimates; the above-mentioned estimate for vaccine effectiveness (VE) against hospitalization is based on a one case only, which is the reason for the wide confidence interval that is compatible with any VE estimate (∞-100%). A hospital-based case-control study from Spain showed that use of several pandemic vaccines was associated with 90% effectiveness in preventing laboratory-confirmed H1N1 infections among hospitalized patients. That study was not population-based and was limited by small number of fully-vaccinated subjects (only 7 subjects received a pandemic vaccine ≥ 7 days before symptom onset).

Two Canadian studies examined the effectiveness of the GSK adjuvanted H1N1 vaccine: one was very small (28 cases) and was limited to children under 10 years. The study by Skowronski et al. that used data from the Canadian VE sentinel network did not examine VE against hospitalization and it, too, was very small.

In the Canadian province of Manitoba, mass immunization against pandemic H1N1 commenced October 26th 2010 using primarily large scale vaccination clinics led by public health teams and lasted approximately 8 weeks. Initially, the Canadian-manufactured Arepanrix®, an AS03-adjuvanted split virion pandemic H1N1 vaccine (GlaxoSmithKline [GSK]), was used to vaccinate adults and children over 6 months of age. Later on, two nonadjuvanted vaccines, from CSL Limited and GSK, were offered to pregnant women and children over 10 years of age. The seasonal trivalent inactivated influenza vaccines (TIV)-Fluviral® (GSK) and Vaxigrip® (Sanofi Pasteur) - were less frequently administered.

All vaccines were offered free of charge, but limited vaccine supply at campaign start necessitated the development of priority groups for early vaccination. The initial priority group in Manitoba included health care workers, Aboriginal persons, pregnant women, 6-60 months-old children, individuals under 65 years with chronic medical conditions, immunocompromised individuals and residents of remote communities. On November 18,2010, the pandemic H1N1 vaccines were made available to the whole population.

This study evaluates the effectiveness of the GSK adjuvanted and non-adjuvanted pH1N1 vaccines used in Manitoba in preventing hospitalization and severe illness. The advantages of the proposed study over the existing literature are related to the availability of high-quality population-based health administrative databases that cover a well-defined population. The whole population of Manitoba is eligible and available for inclusion in the study, so selection bias is not a concern. Ascertainment of cases is virtually complete because all admitted influenza or pneumonia cases in the province are captured by the Hospital Abstract database. The availability of detailed histories of vaccination, through the unique Manitoba Immunization Registry eliminates recall bias, reduces vaccine use measurement errors (e.g., due to patient confusion about what vaccines were received) and permits detailed assessments of the effect of the timing of vaccination on the risk of hospitalization. These detailed analyses will be facilitated by the large sample size (40% of Manitoba's 1.2 million population were vaccinated).

ELIGIBILITY:
Inclusion Criteria:

* Any adult or child > 6 months of age who normally resides in Manitoba and who has been continuously covered during the study period and with a diagnosis of influenza (ICD-10: J09-J11) or pneumonia (ICD-10: J12-J18) will be eligible for inclusion as cases in the study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any adult or child > 6 months of age who normally resides in Manitoba and who has been continuously covered during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1860 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization with laboratory-confirmed influenza or pneumonia | Three months
  Data records of hospitalization with laboratory-confirmed influenza or pneumonia

SECONDARY OUTCOMES:
Hospitalization with influenza or pneumonia | 14 weeks
  Data records of hospitalization with influenza or pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Salah Mahmud, MD, PhD, Principal Investigator — Assistant Professor, University of Manitoba
Locations (1):
- International Centre for Infectious Diseases, Winnipeg, Manitoba, Canada